CLINICAL TRIAL: NCT05883384
Title: Validity of Cow's Milk-related Symptom Score Among Children Suspected to Have Cow's Milk Protein Allergy.
Brief Title: Validity of Cow's Milk-related Symptom Score Among Children Suspected to Have Cow's Milk Protein Alergy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hend Abdelrahim Saber, assistant lecture at pediatric department, Sohag University
Other Study IDs: Soh-Med-23-01-01
Record Dates: First submitted 2023-02-22; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Cow's Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity | interventions — Occult Blood; Blood Cell Count

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with cow milk protein allergy: apply CoMiSS on patient suspected to have cow milk protein allergy.
  Interventions: Other: stool analysis , CBC, specific IgE FOR Cow milk protein allergy

INTERVENTIONS:
Other: stool analysis , CBC, specific IgE FOR Cow milk protein allergy — apply CoMiSS and food challenge test on patient whom suspected to have cow milk protein allergy.

SUMMARY:
Cow's milk protein allergy is a sensitivity reaction against cow's milk protein and and is calcified as IgE-medaited, non- IgE mediated and mixed type according to the underlying immunological mechanism.

Cow's Milk related Symptom Score ( CoMiSS) Considers general manifestation and dermatological, gastrointestinal and respiratory symptoms.

ELIGIBILITY:
Inclusion criteria :

* Age: from birth up to five years...
* Sex: both Males and females
* All children who suspected to have Cow's Milk Allergy that have the following symptoms (chronic unexplained failure to thrive, regurgitation , chronic abdominal distension, skin manifestation such as urticaria & eczema and respiratory symptoms such as chronic cough, recurrent wheezy chest).

Exclusion criteria

* Functional GIT disorders such irritable bowel syndrome , Gastroesophageal reflux disease according to Rome IV criteria in children
* Organic gastrointestinal diseases like coeliac disease , cystic fibrosis.
* Chronic gastrointestinal infections as parasitic infections.

Ages: 1 Minute to 5 Years | Sex: All
Age Groups: Child
Study Population: males and females from birth up to five years who suspected to have Cow's Milk Allergy that have the following symptoms (chronic unexplained failure to thrive, regurgitation , chronic abdominal distension, skin manifestation such as urticaria & eczema and respiratory symptoms such as chronic cough, recurrent wheezy chest).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
patient who are diagnosed as cow milk protein allergy by CoMiss | one year
  measure the accuracy percentage (%) of the Cow's milk-related symptoms score in diagnosis of cow milk allergy at pediatrics department in Sohag hospital university
interpretation of the Cow's milk-related symptoms score | one year
  The scoring ranges from 0 to 33. Each symptom has a maximal score of 6, except respiratory symptoms where the maximal score is 3.
  * If final score > 12, the symptoms are likely cow's milk related. This could potentially be CMPA.
  * If final score < 12, the symptoms are less likely related to cow's milk. Look for other causes.
  * CMPA diagnosis can only be confirmed by an elimination diet followed by an oral food challenge.
Food Challenge Test | one year
  positive or negative Food Challenge Test

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Elieh Ali Komi D, Shafaghat F, Zwiener RD. Immunology of Bee Venom. Clin Rev Allergy Immunol. 2018 Jun;54(3):386-396. doi: 10.1007/s12016-017-8597-4. PMID 28105558
- [Background] Aziz I, Simren M. The overlap between irritable bowel syndrome and organic gastrointestinal diseases. Lancet Gastroenterol Hepatol. 2021 Feb;6(2):139-148. doi: 10.1016/S2468-1253(20)30212-0. Epub 2020 Nov 13. PMID 33189181
- [Background] Schoemaker AA, Sprikkelman AB, Grimshaw KE, Roberts G, Grabenhenrich L, Rosenfeld L, Siegert S, Dubakiene R, Rudzeviciene O, Reche M, Fiandor A, Papadopoulos NG, Malamitsi-Puchner A, Fiocchi A, Dahdah L, Sigurdardottir ST, Clausen M, Stanczyk-Przyluska A, Zeman K, Mills EN, McBride D, Keil T, Beyer K. Incidence and natural history of challenge-proven cow's milk allergy in European children--EuroPrevall birth cohort. Allergy. 2015 Aug;70(8):963-72. doi: 10.1111/all.12630. Epub 2015 May 18. PMID 25864712
- [Background] Vandenplas Y, Mukherjee R, Dupont C, Eigenmann P, Host A, Kuitunen M, Ribes-Koninkx C, Shah N, Szajewska H, von Berg A, Heine RG, Zhao ZY; on behalf the Chinese CoMiSS Investigator Team.. Protocol for the validation of sensitivity and specificity of the Cow's Milk-related Symptom Score (CoMiSS) against open food challenge in a single-blinded, prospective, multicentre trial in infants. BMJ Open. 2018 May 17;8(5):e019968. doi: 10.1136/bmjopen-2017-019968. PMID 29773698